CLINICAL TRIAL: NCT00965601
Title: A Pilot Study on the Use of Nociceptive Flexion Reflex for Fibromyalgia
Acronym: NFR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Dennis C. Ang, MD, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NFR 080554; IU Internally funded
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2009-08

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CTB Group (Active Comparator): Subjects will receive workbook assignments a series of six phone intervention interviews of Cognitive Behavioral Therapy (CBT)
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Usual Care (No Intervention): Subjects will not receive any type of intervention

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Subjects randomized to the Active Arm will receive workbook assignments a series of six phone intervention interviews of Cognitive Behavioral Therapy (CBT)
  Arms: CTB Group

SUMMARY:
The investigators are doing this study to better understand the role of the central nervous system in processing painful stimuli in patients with fibromyalgia. Specifically, the investigators would like to know whether the central nervous system processing of painful stimuli changes with time and with talk therapy. In addition, the investigators are investigating how changes in your fibromyalgia symptoms may affect certain markers or proteins in your blood.

DETAILED DESCRIPTION:
Overall Design

Female patients with FM will be enrolled in this 12-week prospective cohort study. To effect change in patient's symptoms, subjects (n=30) will be randomized to receive six sessions of phone-based cognitive behavioral therapy (CBT) or to 'usual' care. CBT will be provided from week 1 (baseline) to week 6. Outcome assessments (i.e., self-report symptom questionnaires, plasma neuropeptide levels and NFR) will be performed at baseline, week 6 and week 12. Subjects who not complete all three testing phases of the study will be reported as withdraws, and will be replaced as needed until a total of 30 volunteers have completed this study:

Volunteers will be asked to visit the Fibromyalgia Clinical Research Center on 3 different occasions: baseline (Screening), week 6, and week 12.

During the first visit subjects will be randomly assigned to one of two groups. Similar to flipping a coin, you have a 50% chance of being assigned to either one of two groups: a) telephone-based educational instruction group or b) usual care group. Subjects who are randomly assigned to educational instruction group will receive one phone call per week for the first six weeks of the study. During the phone conversation, you will receive instructions in managing your pain. If subjects are assigned to the educational instruction group, subjects must agree to allow us to audiotape the telephone conversation. Audio-taping the telephone conversations will help us give you the highest quality of instruction. On the other hand, subjects assigned to the usual care group will receive no telephone calls from the research team.

During each visit subjects will be asked to do the following:

1. Complete a comprehensive questionnaire (computer-based or the traditional paper and pen format) in regard to how fibromyalgia affects your daily living.

   Risks: You may feel uncomfortable or care not to answer a particular question. To minimize these risks, you can tell the researcher that you feel uncomfortable or do not wish to answer the question.
2. Provide a blood sample (10 ml).The purpose or this blood test is to examine changes in certain blood markers in relation to your changes in your symptoms

   Risks: The physical risks associated with participation in this study are with the blood draw. The process of drawing blood may cause bleeding, bruising, pain, lightheadedness, and some minor swelling around the area of the needle stick. Occasionally an infection or bleeding may develop where the needle was placed in the vein. To minimize these risks, the blood specimen will be obtained by experienced technicians.
3. Undergo nociceptive flexion reflex (NFR) testing. This test examines how your body responds to painful stimuli. To begin each testing session, electrodes used to measure the nociceptive flexion reflex will be attached to your left leg. To measure the reflex, we will administer a series of electrical stimuli to the ankle of your left foot. After each stimulus you will be asked to rate the stimulus intensity using a scale with anchors of 0 (no sensation), 50 (pain threshold), and 100 (maximum tolerable). This procedure is used to determine the intensity of stimulus required to elicit a nociceptive flexion reflex response from your left hamstring muscle. This reflex is so small that you may not even notice any activity in your leg muscles. The intensity of electrical stimuli will be increased slowly until a reflex response is shown, but the intensity will NEVER exceed that which you rate as a "100" (maximum tolerable). At the higher intensities, the electrical stimulus is described by others as feeling like a "brief pinprick" or "carpet shock".

We will use the same procedure to assess your pain tolerance threshold for electrical stimulation to your ankle. Stimulus intensity will be increased slowly and you will be asked to rate each stimulus on the 0-100 scale. The procedure will end as soon as you provide a stimulus intensity rating of "100" (maximum tolerable).

Risks: The nociceptive flexion reflex procedure is likely to elicit temporary discomfort, increases in heart rate and blood pressure as well as sensations of discomfort or pain. Further, preparation of the skin required to apply electrodes may be mildly irritating or uncomfortable, and may leave behind some redness of the skin that could require a few days to heal. To minimize these risks, only well trained technicians will conduct this test. It is important to note that this test is similar to an EMG (electromyogram) study - a test commonly done in routine medical care.

ELIGIBILITY:
Inclusion Criteria:

* 1. Female volunteers who have been diagnosed with fibromyalgia by a rheumatologist.
* 2. Overall body pain average score ≥ 4
* 3. Age range: 18 to 65 years old
* 4. You must be on stable doses of anyone of these fibromyalgia-related medications for at least 4 weeks: cyclobenzaprine, tramadol, gabapentin, pregabalin, amitriptyline, nortriptyline, trazodone, sertraline, fluoxetine, paxil, remeron, venlafaxine and duloxetine.
* 5. Willingness to restrict any change (add or switch or change in the dose) of any fibromyalgia-related medication for 12 weeks.

Exclusion Criteria:

* 1. Volunteers who have long-standing history of diabetes (> 2 years), or have been diagnosed with any type of peripheral neuropathy.
* 2. Have a prior history of myocardial infarction (heart attack) or unstable angina or other heart arrhythmias.
* 3. Have been diagnosed with multiple sclerosis or any other demyelinating disorder.
* 4. Have planned to undergo an elective surgery over the next 12 weeks.
* 5. Have other major rheumatic conditions (i.e. rheumatoid arthritis, systemic lupus erythematosus, scleroderma and other connective tissue disease)
* 6. Are currently pregnant or actively trying to become pregnant

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Aim 1: Test the feasibility and subject acceptability of a potentially objective tool (NFR) for measuring pain severity. | Baseline, Week 9, and Week 12

SECONDARY OUTCOMES:
Aim 2: Determine the longitudinal relationships of changes in patients' symptoms with changes in plasma levels of neuropeptides and NFR pain threshold. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dennis C Ang, MD, Principal Investigator — Indiana University Department of Medicine
Locations (1):
- National Institute of Fitness and Sport; IUPUI Campus, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Ang DC, Chakr R, Mazzuca S, France CR, Steiner J, Stump T. Cognitive-behavioral therapy attenuates nociceptive responding in patients with fibromyalgia: a pilot study. Arthritis Care Res (Hoboken). 2010 May;62(5):618-23. doi: 10.1002/acr.20119. PMID 20191481